CLINICAL TRIAL: NCT00799643
Title: Targeting Inflammation in Type 2 Diabetes: Clinical Trial Using Salsalate
Brief Title: Targeting Inflammation Using Salsalate for Type 2 Diabetes-Stage II
Acronym: TINSALT2D-II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS 06-20-2; U01DK074556 (NIH)
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus (T2D); Inflammation; Obesity; Metabolic Syndrome; Salicylates
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Obesity; Metabolic Syndrome | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Salsalate, 3.5 g/d orally, divided dosing
  Interventions: Drug: Salsalate
- 2 (Placebo Comparator): Salsalate Placebo, orally, divided dosing
  Interventions: Drug: Salsalate Placebo

INTERVENTIONS:
Drug: Salsalate — Salsalate 3.5 g/d orally, divided dosing
  Other Names: disalsid
  Arms: 1
Drug: Salsalate Placebo
  Arms: 2

SUMMARY:
Growing evidence over recent years supports a potential role for low grade chronic inflammation in the pathogenesis of insulin resistance and type 2 diabetes. In this study we will determine whether salsalate, a member of the commonly used Non-Steroidal Anti-Inflammatory Drug (NSAID) class, is effective in lowering sugars in patients with type 2 diabetes. The study will determine whether salicylates represent a new pharmacological option for diabetes management. The study is conducted in two stages. Enrollment in the first stage is complete. The primary objective of the first stage was to select a dose of salsalate that is both well-tolerated and demonstrates a trend toward improvement in glycemic control. The primary objective of Stage 2 of the study is to evaluate the effects of salsalate on blood sugar control in diabetes; the tolerability of salsalate use in patients with type 2 diabetes (T2D); and the effects of salsalate on measures of inflammation, the metabolic syndrome, and cardiac risk.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes on diet and exercise therapy or monotherapy with metformin, insulin secretagogue (including SFU, non-SFU, and dipeptidyl peptidase IV (DPP-4) inhibitors), alpha-glucosidase inhibitors, or bile acid sequestrants (dosed once per day such that study drug can be administered ≥ 4 hours prior to sequestrant); or a combination of up to two of these at maximal dose. Dosing must be stable for 8 weeks prior to screening. Participant must have been diagnosed with T2D at least 8 weeks before screening.
2. FPG ≤ 225 mg/dL and HbA1c≥7% and ≤ 9.5% at screening.
3. Age ≥18 and <75
4. Women of childbearing potential agree to use an appropriate contraceptive method (hormonal, IUD, or diaphragm)

Exclusion Criteria:

1. No prior participation in Stage I of TINSAL-T2D ; exception: a participant who failed screening for HbA1c in Stage I will be allowed to re-screen for Stage II.
2. Type 1 diabetes and/or history of ketoacidosis determined by medical history
3. History of severe diabetic neuropathy including autonomic neuropathy, gastroparesis or lower limb ulceration or amputation
4. History of long-term therapy with insulin (>30 days) within the last year
5. Therapy with rosiglitazone (Avandia) or pioglitazone (Actos), alone or in combination in the previous 6 months; or exendin-4 (Byetta), alone or in combination in the previous 3 months
6. Pregnancy or lactation
7. Patients requiring oral corticosteroids within 3 months or recurrent continuous oral corticosteroid treatment (more than 2 weeks)
8. Use of weight loss drugs [e.g., Xenical (orlistat), Meridia (sibutramine), Acutrim (phenylpropanol-amine), or similar over-the-counter medications] within 3 months of screening or intentional weight loss of ≥ 10 lbs in the previous 6 months
9. Surgery within 30 days prior to screening
10. Serum creatinine >1.4 for women and >1.5 for men or eGFR <60 [possible chronic kidney disease stage 3 or greater calculated using the Modification of Diet in Renal Disease (MDRD) equation
11. History of chronic liver disease including hepatitis B or C
12. History of peptic ulcer or endoscopy demonstrated gastritis
13. History of acquired immune deficiency syndrome or human immunodeficiency virus (HIV)
14. History of malignancy, except participants who have been disease-free for greater than 10 years, or whose only malignancy has been basal or squamous cell skin carcinoma
15. New York Heart Association Class III or IV cardiac status or hospitalization for congestive heart failure
16. History of unstable angina, myocardial infarction, cerebrovascular accident, transient ischemic attack or any revascularization within 6 months
17. Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg on three or more assessments on more than one day). If on blood pressure medications, dosing should be stable for 2 weeks prior to randomization.
18. History of drug or alcohol abuse, or current weekly alcohol consumption >10 units/week (1 unit = 1 beer, 1 glass of wine, 1 mixed DCCktail containing 1 ounce of alcohol)
19. Hemoglobin <12 g/dL (males), <10 g/dL (females) at screening*
20. Platelets <100,000 cu mm at screening
21. AST (SGOT) >2.50 x ULN or ALT (SGPT) >2.50 x ULN at screening
22. Total Bilirubin >1.50 x ULN at screening
23. Triglycerides (TG) >500 mg/dL at screening
24. Poor mental function or any other reason to expect patient difficulty in complying with the requirements of the study
25. Previous allergy to aspirin
26. Chronic or continuous use (daily for more than 7 days) of nonsteroidal anti-inflammatory drugs within the preceding 2 months
27. Use of warfarin (Coumadin), clopidogrel (Plavix), dipyridamole (Persantine), heparin or other anticoagulants
28. Use of probenecid (Benemid, probalan), sulfinpyrazone (Anturane) or other uricosuric agents
29. Macroalbuminuria, defined as spot urine protein >300 mcg/mg Cr at screening
30. Pre-existing chronic tinnitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Shoelson, MD, PhD, Principal Investigator — Joslin Diabetes Center; Allison B. Goldfine, MD, Study Director — Joslin Diabetes Center; Vivian Fonseca, MD, Study Director — Tulane University; Kathleen Jablonski, PhD, Study Director — George Washington University; Myrlene Staten, MD, Study Director — National Institute of Diabetes & Digestive & Kidney Diseases (NIDDK)
Locations (21):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Chapel Medical Group, New Haven, Connecticut
  - Emory University School of Medicine, Atlanta, Georgia
  - Kaiser Permanente, Tucker, Georgia
  - Indiana University, Indianapolis, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Medstar Research Institute, Hyattsville, Maryland
  - Dr. Rudo, Westminster, MD, Westminster, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Columbia University, New York, New York
  - Lang Medical Center, Queens, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Carolina's Health Care, Charlotte, North Carolina
  - University of North Carolina, Durham, North Carolina
  - University of Texas Southwestern, Dallas, Texas
  - Scott and White, Temple, Texas

REFERENCES:
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Pyle L, Staten MA, Shoelson SE; TINSAL-T2D (Targeting Inflammation Using Salsalate in Type 2 Diabetes) Study Team. The effects of salsalate on glycemic control in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2010 Mar 16;152(6):346-57. doi: 10.7326/0003-4819-152-6-201003160-00004. PMID 20231565
- [Result] Goldfine AB, Fonseca V, Jablonski KA, Chen YD, Tipton L, Staten MA, Shoelson SE; Targeting Inflammation Using Salsalate in Type 2 Diabetes Study Team. Salicylate (salsalate) in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2013 Jul 2;159(1):1-12. doi: 10.7326/0003-4819-159-1-201307020-00003. PMID 23817699
- [Derived] Goldfine AB, Buck JS, Desouza C, Fonseca V, Chen YD, Shoelson SE, Jablonski KA, Creager MA; TINSAL-FMD (Targeting Inflammation Using Salsalate in Type 2 Diabetes-Flow-Mediated Dilation) Ancillary Study Team. Targeting inflammation using salsalate in patients with type 2 diabetes: effects on flow-mediated dilation (TINSAL-FMD). Diabetes Care. 2013 Dec;36(12):4132-9. doi: 10.2337/dc13-0859. Epub 2013 Oct 15. PMID 24130358
- See also: description of trial for patients and medical professionals — http://tinsalt2d.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Enrollment number in the protocol section (638) is higher than the number of participants Started in the Participant Flow module (286) due to screen failures and drop out prior to randomization.
Groups:
- Placebo: Placebo for salsalate, orally, divided dosing
- Salsalate: Salsalate, 3.5 g/d orally,divided dosing
Period: Overall Study
Arm/Group | Placebo | Salsalate
Started | 140 | 146
Completed | 115 | 119
Not Completed | 25 | 27

BASELINE CHARACTERISTICS:
Groups:
- Salsalate: Salsalate, 3.5 g/d orally, divided dosing
- Total: Total of all reporting groups
Arm/Group | Placebo | Salsalate | Total
Number analyzed (Participants) | 140 | 146 | 286
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 118 | 230
  >=65 years | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (10) | 55.8 (9.2) | 55.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 129
  Male | 75 | 82 | 157
Region of Enrollment [Number; unit: participants]
  United States | 140 | 146 | 286

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome for the TINSAL-T2D Study is Change in HbA1c Level From Baseline to Week 48 From Baseline, Compared Between Treatment Groups.
Description: HbA1c (%, percentage of HbA1c) change from baseline.
Time Frame: 48 weeks from baseline
Population: Participants with complete data at both Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: HbA1c units are %
Arm/Group | Placebo | Salsalate
Number analyzed (Participants) | 137 | 146
HbA1c units are % | -0.04 [-0.07 to 0.15] | -0.33 [-0.44 to -0.22]

2. Secondary Outcome: Change From Baseline in Fasting Glucose Over Time.
Time Frame: 48 weeks from baseline
Population: Participants with complete data at both Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Placebo | Salsalate
Number analyzed (Participants) | 137 | 146
mg/dl | 2.0 [-1.9 to 5.9] | -13.1 [-16.9 to -9.2]

3. Secondary Outcome: Response Rates for Reduction in Fasting Glucose of ≥20 mg/dl, a Reduction in HbA1c of ≥0.5%, and a Reduction in HbA1c of ≥0.8%
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change in Lipids (Low-density Lipoprotein Cholesterol [LDL-C], Non-high-density Lipoprotein Cholesterol [Non-HDL-C], Triglycerides [TG], Total Cholesterol [TC], High-density Lipoprotein Cholesterol [HDL C], TC/HDL-C Ratio, and LDL-C/HDL-C Ratio)
Time Frame: 48 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Changes in WBC and Differential, High-sensitivity C Reactive Protein (hsCRP), Other Inflammatory Markers
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Response Rates for Exceeding Hyperglycemic Targets Between Active and Placebo Treated Groups; Need for Rescue Therapy; Need for Discontinuation of Study Medication
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Response Rates in Patients Initially Treated With Lifestyle Modification, Insulin Secretagogue, Metformin or Combination Therapy
Time Frame: 24 and 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Placebo | Salsalate
Serious Adverse Events (participants affected / at risk) | 6/140 | 10/146
Other Adverse Events (participants affected / at risk) | 64/140 | 85/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=140) | Salsalate (N=146)
Hematuria/Bladder Cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostate Hypertrophy/TURP (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic Lymphoid Leukemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gallstones/Cholycystectomy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 2 (2)
Reactive Airway Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Traumatic Fracture or Joint Diastasis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cervical Disectomy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | Salsalate (N=146)
Tinnitus (Ear and labyrinth disorders) | 7 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 20
Vomiting (Gastrointestinal disorders) | 10 | 11
Muscle Stiffness (Musculoskeletal and connective tissue disorders) | 9 | 14
Dizzy (General disorders) | 10 | 11
Weakness or Fatigue (General disorders) | 9 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No